CLINICAL TRIAL: NCT03810794
Title: Clinical Evaluation on the Therapeutic Effect of Acupuncture Treatment for Alzheimer's Disease: Multicenter Randomized Controlled Trial
Brief Title: Clinical Evaluation on the Therapeutic Effect of Acupuncture Treatment for Alzheimer's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jian Pei,MD (Other)
Collaborators: Shanghai Mental Health Center (Other); Huashan Hospital (Other)
Responsible Party: Sponsor-Investigator, Jian Pei,MD, Department Chief, Shanghai University of Traditional Chinese Medicine
Organization: Shanghai University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18401970500
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease; Cognitive Impairment
Keywords: Acupuncture Treatment; Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Acupuncture Therapy; Donepezil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupuncture Treatment Group (Experimental): Participants in this group will be given acupuncture treatment in combination with donepezil for 12 weeks.
  Interventions: Other: Acupuncture; Drug: Donepezil
- Donepezil Group (Active Comparator): Participants in this group will be given only donepezil for 12 weeks.
  Interventions: Drug: Donepezil

INTERVENTIONS:
Other: Acupuncture — The main acupoints are DU 24, EX-HN 3, DU 20, EX-HN 1, GB 12, HT 7, KI 6, GB39, and then selecting other acupoints according to TCM syndrome. The electric stimulator will be applied to DU 24, GB 12, HT 7, and LR 3 or SP 6 with a disperse-dense wave of 2/50 Hz, 0.5-1.0 mA. There are three sessions per week with each session lasting for 30 min. There will be 12 weeks of treatment for each participant in total.
  Arms: Acupuncture Treatment Group
Drug: Donepezil — Donepezil 5 mg will be given once daily before bed-time for 12 weeks. After the clinical trial, participants will be given conventional treatment clinically.
  Other Names: Donepezil Hydrochloride Tablets

SUMMARY:
The objective of this proposed study is to evaluate the effect and safety of acupuncture combined therapy on cognitive function, daily living ability and quality of life of Alzheimer's disease by using the international dementia certification scale. In this 12-week, assessor-blind, a Multi-center randomized, controlled study of acupuncture as additional treatment with Donepezil, a total of 180 patients with Alzheimer's disease will be recruited. The patients will be randomly assigned to acupuncture combined with Donepezil (n =90) or Donepezil treatment (n =90). (36 sessions, 3 sessions a week). Changes in the cognition over time measured using ADAS-cog is the primary outcome. MMSE, ADCS-ADL and QOL-AD are the secondary outcomes. The study will be conducted at LongHua Hospital Shanghai University of Traditional Chinese Medicine, Huashan Hospital Fudan University, and Mental Health Center Shanghai Jiao Tong University School of Medicine.

DETAILED DESCRIPTION:
Objective: To evaluate the effect and safety of acupuncture combined therapy on cognitive function, daily living ability and quality of life of Alzheimer's disease by using the international dementia certification scale.

Methods/design: A total of 180 participants with mild to moderate Alzheimer's disease will be randomly assigned to either an acupuncture combined with donepezil group or a donepezil group with a ratio of 1:1. Participants in the acupuncture combined with donepezil group will receive acupuncture treatment in combination with donepezil for 12 weeks and at same time taking donepezil. The main acupoints are DU 24, EX-HN 3, DU 20, EX-HN 1, GB 12, HT 7, KI 6, GB39, and then selecting other acupoints according to TCM syndrome. The electric stimulator will be applied to DU 24, GB 12, HT 7, and LR 3 or SP 6 with a disperse-dense wave of 2/50 Hz, 0.5-1.0 mA. There are 3 sessions per week with each session lasting for 30 min. There will be 12 weeks of treatment for each participant in total. Donepezil 5 mg will be given once daily before bed-time for 12 weeks. After the clinical trial, participants will be given conventional treatment clinically. Participants in the control group will take donepezil only. A follow-up will be conducted 24 weeks after the treatment. The primary outcome is the change and effective rate from baseline in the ADAS-cog score measured at week 12. The secondary outcomes contains The change from baseline in MMSE score, ADCS-ADL score, QOL-AD score measured at weeks 12, 24 and 36.

ELIGIBILITY:
Inclusion Criteria:

* aged between 50-85 years
* the diagnostic criteria of Neurological Communicative Disorders and Stroke and the Alzheimer Disease and Related Disorders Association (NINCDS-ADRDA)
* cognitive impairment based on the scores of the Chinese version of the Mini Mental State Examination (MMSE) (patients with mild to moderate Alzheimers disease, 11≤primary school degree≤22, 11≤junior high school degree or above≤26
* magnetic resonance imaging (MRI) confirmation of atrophy of the hippocampus or the medial temporal lobe volume, MRI manifestation of high possibility of Alzheimer Disease
* the Medial Temporal Lobe Atrophy Rating Scale (MTA-scale) score (≥2 for those under 75 years, and ≥3 for those over 75 years)
* voluntarily joining this study with informed consents

Exclusion Criteria:

* cognitive impairment caused by other factors (e.g. vascular dementia, dementia with Lewy bodies, frontotemporal dementia, hormone or metabolic abnormalities, hypothyroidism, folic acid or vitamin B12 deficiency, delirium or other mental and emotional disorders (such as schizophrenia and depression))
* a serious heart condition, hepatic disease, renal system disease, hematopoietic system disease, or whole-body malnutrition
* aphasia, disturbance of consciousness, or failure to cooperate with the related examinations due to physical disability
* anticoagulant treatments such as warfarin or heparin
* use of pacemakers or receiving acupuncture in the past 2 weeks

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-cognition(ADAS-cog) | Baseline(week -2), treatment at week 12
  The primary outcome are the change and effective rate from baseline in the Alzheimer's Disease Assessment Scale-cognition(ADAS-cog) score measured at week 12. The maximum score of the ADAS-cog is 70 including 12 items. The questions in this scale contain word recall task, naming objects and fingers, following commands, constructional praxis, ideational praxis, orientation, word recognition task, remembering test directions, spoken language, word-finding difficulty, comprehension and attention. In general, a normal score for someone who does not have AD or another type of dementia is 5. The higher scores indicate higher degree of cognitive dysfunction.

SECONDARY OUTCOMES:
Minimum Mental State Examination(MMSE) | Baseline(week -2), Treatment at week 12, Follow-up at weeks 12 and 24.
  The change from baseline in total Minimum Mental State Examination(MMSE) score should be measured at weeks 12, 24 and 36. The maximum score of the MMSE is 30. The questions in this scale include orientation to time, orientation to place, attention and calculation, recall of three words, and visual construction. The lower scores indicate higher degree of cognitive dysfunction. The score is related to degree of education. In general, the score of normal people is 27-30.
Alzheimer's Disease Cooperative Study-Activity of Daily Living(ADCS-ADL) | Baseline(week -2), Treatment at week 12, Follow-up at weeks 12 and 24.
  The change from baseline in the Alzheimer's Disease Cooperative Study-Activity of Daily Living(ADCS-ADL) score should be measured at weeks 12, 24 and 36. The maximum of the ADCS-ADL score is 54 containing 19 domains about assessment of basic and operational ability of daily living. The higher scores indicate higher ability of daily living.
Quality of Life-Alzheimer's Disease(QOL-AD) | Baseline(week -2), Treatment at week 12, Follow-up at weeks 12 and 24.
  The change from baseline in the Quality of Life-Alzheimer's Disease(QOL-AD) score should be measured at weeks 12, 24 and 36. The QOL-AD score includes 13 items about physical health, mental health, social and financial assessment, and quality of life. The total score ranges from 13 to 52. The higher scores indicate higher quality of life.
fractional amplitude of low frequency fluctuation (fALFF) | Baseline(week -2), Treatment at week 12
  fALFF aquired by fMRI technique measures the relative contribution of low frequency fluctuations within a speciﬁc frequency band to the whole detectable frequency range
functional connectivity (FC) | Baseline(week -2), Treatment at week 12
  FC aquired by fMRI technique measures the functional connectivity of specific brain regions to the whole brain

CONTACTS AND LOCATIONS:
Overall Officials: Jian Pei, Doctor, Study Chair — Shanghai University of Traditional Chinese Medicine; Houguang Zhou, Doctor, Study Director — Huashan Hospital; Tao Wang, Doctor, Study Director — Mental Health Center Shanghai Jiao Tong University School of Medicine
Locations (3):
- China (3):
  - LongHua Hospital Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Shanghai Mental Center, Shanghai Jiaotong University of Medicial School, Shanghai, Shanghai Municipality
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Fu QH, Pei J, Zhou HG, Wang T, Zhan YJ, Tao L, Xu J, Zhou Q, Wang LY. Effect of acupuncture with donepezil based on syndrome differentiation on cognitive function in patients with mild-to-moderate Alzheimer's disease: a study protocol for a multicenter randomized controlled trial. Trials. 2022 Aug 19;23(1):695. doi: 10.1186/s13063-022-06532-1. PMID 35986297
- [Derived] Zhan Y, Fu Q, Pei J, Fan M, Yu Q, Guo M, Zhou H, Wang T, Wang L, Chen Y. Modulation of Brain Activity and Functional Connectivity by Acupuncture Combined With Donepezil on Mild-to-Moderate Alzheimer's Disease: A Neuroimaging Pilot Study. Front Neurol. 2022 Jul 11;13:912923. doi: 10.3389/fneur.2022.912923. eCollection 2022. PMID 35899271